CLINICAL TRIAL: NCT00562120
Title: A Randomized, Double Blind, Double Dummy, Placebo Controlled, Four Way Crossover Study To Determine The Effects Of An H3 Receptor Antagonist (PF-03654746) On Congestion Following A Nasal Allergen Challenge In Subjects With Seasonal Allergic Rhinitis.
Brief Title: A Study to Test a New Decongestant in Patients With Allergic Rhinitis Following a Nasal Allergen Challenge
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A8801003
Record Dates: First submitted 2007-11-19; First posted 2007-11-21 (Estimated); Results first posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — fexofenadine; N-ethyl-3-fluoro-3-(3-fluoro-4-(pyrrolidinylmethyl)phenyl)cyclobutanecarboxamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Allegra (Active Comparator)
  Interventions: Drug: Allegra
- Allegra-D (Active Comparator)
  Interventions: Drug: Allegra-D
- PF-03654746 (Experimental)
  Interventions: Drug: PF-03654746

INTERVENTIONS:
Drug: Placebo — A single oral dose of Placebo is dosed during the study in order to ascertain the effect of placebo on measures and in order to maintain the blind of the other drugs.
  Arms: Placebo
Drug: Allegra — A single oral dose of Allegra is dosed to subjects in combination with PF-03654746.
  Arms: Allegra
Drug: Allegra-D — A single oral dose of Allegra-D is dosed to subjects as an active comparator.
  Arms: Allegra-D
Drug: PF-03654746 — A single oral dose of PF-03654746 is the investigational drug being studied.
  Arms: PF-03654746

SUMMARY:
An H3 receptor antagonist should reduce the congestion associated with allergic rhinitis. A nasal allergen challenge will be given to patients to induce rhinitis symptoms and acoustic rhinometry will be used to measure the congestion.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects 19-55 years with allergic rhinitis requiring treatment within the previous 2 years.
* Subjects that respond to a ragweed nasal allergen challenge at screening.

Exclusion Criteria:

* History of asthma or FEV1 < 80% predicted.
* Significant concomitant disease or medications.
* Symptoms of allergic rhinitis within 2 weeks prior to screening.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2007-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Omaha, Nebraska, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A8801003&StudyName=A%20study%20to%20test%20a%20new%20decongestant%20in%20patients%20with%20allergic%20rhinitis%20following%20a%20nasal%20allergen%20challenge

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D: PF-03654746 10 milligram (mg) capsule and Allegra (fexofenadine 60 mg) tablet-in-capsule along with placebo matched to Allegra-D (fexofenadine 60 mg in combination with pseudoephedrine 120 mg) tablet-in-capsule on Day 1 in the first intervention period; followed by placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the second intervention period; then PF-03654746 1 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the third intervention period; and placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with Allegra-D tablet-in-capsule on Day 1 in the fourth intervention period. A washout period of at least 14 days was maintained between each treatment period.
- PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo: PF-03654746 1 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the first intervention period; followed by PF-03654746 10 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the second intervention period; then placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule and Allegra-D tablet-in-capsule on Day 1 in the third intervention period; and placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with Allegra-D tablet-in-capsule on Day 1 in the fourth intervention period. A washout period of at least 14 days was maintained between each treatment period.
- Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg: Placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with Allegra-D tablet-in-capsule on Day 1 in the first intervention period; followed by PF-03654746 1 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the second intervention period; then placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the third intervention period; and PF-03654746 10 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the fourth intervention period. A washout period of at least 14 days was maintained between each treatment period.
- Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg: Placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the first intervention period; followed by placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with Allegra-D tablet-in-capsule on Day 1 in the second intervention period; then PF-03654746 10 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the third intervention period; and PF-03654746 1 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 in the fourth intervention period. A washout period of at least 14 days was maintained between each treatment period.
Period: First Intervention Period
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 6 | 5 | 5 | 5
Treated | 5 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Randomized but not Treated | 1 | 0 | 0 | 0
Period: Washout Period 1 (At Least 14 Days)
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention Period
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (At Least 14 Days)
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Third Intervention Period
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 3 (At Least 14 Days)
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0
Period: Fourth Intervention Period
Arm/Group | PF-03654746 10 mg, Placebo, PF-03654746 1 mg, Allegra-D | PF-03654746 1 mg, PF-03654746 10 mg, Allegra-D, Placebo | Allegra-D, PF-03654746 1 mg, Placebo, PF-03654746 10 mg | Placebo, Allegra-D, PF-03654746 10 mg, PF-03654746 1 mg
Started | 4 | 5 | 5 | 5
Completed | 4 | 5 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomized at baseline and who received at least 1 dose of double-blind treatment.
Groups:
- Entire Study Population: All participants randomized to any treatment (PF-03654746 10 mg capsule first, PF-03654746 1 mg capsule first, Allegra-D tablet-in-capsule first and placebo first).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 20
Age, Customized [Number; unit: participants]
  18 to 44 years | 15
  45 to 64 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Minimum Cross-Sectional Area (Amin) Proportion Measured Using Acoustic Rhinometry
Description: Acoustic rhinometry: a technique intended for assessment of the geometry of nasal cavity and nasopharynx and for evaluating nasal obstruction. At each time point, there were 2 acoustic rhinometry measurements taken, one for each nostril. Mean of the left and right nostril measurements was taken as measurement at each time point. Minimum Cross-Sectional Area (Amin) at Baseline was defined as mean of 3, 'post-diluent, pre-allergen challenge' measures for each intervention period at 2 hours (hrs) 10 minutes (min), 2 hrs 25 min and 2 hrs 40 min post PF-03654746/placebo dose. Amin 'post-allergen challenge' measures recorded at 2 hrs 55 min, 3 hrs 10 min and 3 hrs 25 min post PF-03654746/placebo dose for each intervention period was averaged to derive single 'post-allergen challenge' value. Amin proportion was defined as ratio of 'post-allergen challenge' value and 'Baseline/pre-allergen challenge value'. Diluent used was saline and allergen was short ragweed extract.
Time Frame: 2 hrs 10 min, 2 hrs 25 min, 2 hrs 40 min post dose (Baseline); 2 hrs 55 min, 3 hrs 10 min, 3 hrs 25 min post dose on Day 1 of each intervention period
Population: Full analysis set included all participants randomized at baseline and who received at least 1 dose of double-blind treatment.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- PF-03654746 10 mg: PF-03654746 10 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 of any of the intervention periods.
- PF-03654746 1 mg: PF-03654746 1 mg capsule and Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 of any of the intervention periods.
- Allegra-D: Placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with Allegra-D tablet-in-capsule on Day 1 of any of the intervention periods.
- Placebo: Placebo matched to PF-03654746 capsule and placebo matched to Allegra tablet-in-capsule along with placebo matched to Allegra-D tablet-in-capsule on Day 1 of any of the intervention periods.
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Number analyzed (Participants) | 20 | 19 | 19 | 19
ratio | 0.760 (0.1504) | 0.742 (0.2552) | 0.717 (0.1935) | 0.795 (0.3044)
Statistical Analysis 1: Comparison: PF-03654746 10 mg vs Placebo; An analysis of variance (ANOVA) mixed model was assessed with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.302, ANOVA — P-value was based on one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 2: Comparison: Allegra-D vs Placebo; An ANOVA mixed model was assessed with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.134, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 3: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.229, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 4: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.544, ANOVA — P-value was based on two-sided test which was underpowered and presented for descriptive purposes only. There were no further adjustments for multiplicity
Statistical Analysis 5: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.710, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.816, ANOVA — [p-value comment as in outcome 1, analysis 4]

2. Primary Outcome: Nasal Volume Proportion Measured Using Acoustic Rhinometry
Description: Acoustic rhinometry: a technique intended for assessment of the geometry of nasal cavity and nasopharynx and for evaluating nasal obstruction. At each time point, there were 2 acoustic rhinometry measurements taken, one for each nostril. Mean of the left and right nostril measurements was taken as measurement at each time point. Nasal volume at Baseline was defined as mean of 3, 'post-diluent, pre-allergen challenge' measures for each intervention period at 2 hrs 10 min, 2 hrs 25 min and 2 hrs 40 min post PF-03654746/placebo dose. Nasal volume 'post-allergen challenge' measures recorded at 2 hrs 55 min, 3 hrs 10 min and 3 hrs 25 min post PF-03654746/placebo dose for each intervention period was averaged to derive single 'post-allergen challenge' value. Nasal volume proportion was defined as ratio of 'post-allergen challenge' value and 'Baseline/pre-allergen challenge value'. Diluent used was saline and allergen was short ragweed extract.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Number analyzed (Participants) | 20 | 19 | 19 | 19
ratio | 0.800 (0.1825) | 0.796 (0.2641) | 0.744 (0.1594) | 0.856 (0.3859)
Statistical Analysis 1: Comparison: PF-03654746 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.269, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 2: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.097, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 3: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.252, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 4: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.479, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.521, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.952, ANOVA — [p-value comment as in outcome 1, analysis 4]

3. Secondary Outcome: Minimum Cross-Sectional Area (Amin) Maximum Fall Measured Using Acoustic Rhinometry
Description: Acoustic rhinometry: a technique intended for assessment of the geometry of the nasal cavity and nasopharynx and for evaluating nasal obstruction. At each time point, there were 2 acoustic rhinometry measurements taken, one for each nostril. The mean of the left and right nostril measurements was taken as the measurement at each time point. Minimum Cross-Sectional Area (Amin) at Baseline was defined as mean of the 3, 'post-diluent, pre-allergen challenge' measures for each intervention period at 2 hrs 10 min, 2 hrs 25 min and 2 hrs 40 min post PF-03654746/placebo dose. Amin 'post-allergen challenge' measures were recorded at 2 hrs 55 min, 3 hrs 10 min and 3 hrs 25 min post PF-03654746/placebo dose for each intervention period. The maximum fall in Amin was calculated as baseline measure minus smallest 'post-allergen challenge' Amin measurement of the 3 measures.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: square centimeter (cm^2)
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Number analyzed (Participants) | 20 | 19 | 19 | 19
square centimeter (cm^2) | 0.155 (0.0876) | 0.157 (0.1159) | 0.204 (0.0951) | 0.190 (0.1510)
Statistical Analysis 1: Comparison: PF-03654746 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.130, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 2: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.663, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 3: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.138, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 4: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.124, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.134, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.978, ANOVA — [p-value comment as in outcome 1, analysis 4]

4. Secondary Outcome: Nasal Volume Maximum Fall Measured Using Acoustic Rhinometry
Description: Acoustic rhinometry: a technique intended for assessment of the geometry of the nasal cavity and nasopharynx and for evaluating nasal obstruction. At each time point, there were 2 acoustic rhinometry measurements taken, one for each nostril. The mean of the left and right nostril measurements was taken as the measurement at each time point. Nasal volume at Baseline was defined as mean of the 3, 'post-diluent, pre-allergen challenge' measures for each intervention period at 2 hrs 10 min, 2 hrs 25 min and 2 hrs 40 min post PF-03654746/placebo dose. Nasal volume 'post-allergen challenge' measures were recorded at 2 hrs 55 min, 3 hrs 10 min and 3 hrs 25 min post PF-03654746/placebo dose for each intervention period. The maximum fall for nasal volume was calculated as baseline measure minus smallest 'post-allergen challenge' nasal volume measurement among the 3 measures.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cubic centimeter (cm^3)
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Number analyzed (Participants) | 20 | 19 | 19 | 19
cubic centimeter (cm^3) | 3.132 (2.4120) | 3.244 (2.3676) | 4.443 (2.9502) | 3.275 (2.7001)
Statistical Analysis 1: Comparison: PF-03654746 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.357, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 2: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.952, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 3: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.480, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 4: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.043, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.087, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.753, ANOVA — [p-value comment as in outcome 1, analysis 4]

5. Secondary Outcome: Nasal Symptom Scores: Nasal Congestion, Nasal Itching, Rhinorrhea
Description: Nasal symptoms included; nasal congestion: participants rated sensation of nasal blockage on 0 (no blockage) to 5 (total blockage) scale, nasal itching: participants rated sensation of nasal itch on 0 (no itch) to 5 (very itchy) scale, rhinorrhea: participants rated sensation of runny nose on 0 (no running) to 5 (very runny) scale. Symptom scores were assessed as mean of each intervention period at specified time-points for 'post-diluent, pre-allergen challenge' measure and 'post-challenge' measure. Post-diluent, pre-allergen challenge (for congestion, itching, rhinorrhea) included 2 hrs 10 min, 2 hrs 25 min and 2 hrs 40 min post PF-03654746/placebo dose at each intervention period and post-allergen challenge (for congestion, itching, rhinorrhea) included 2 hrs 55 min, 3 hrs 10 min and 3 hrs 25 min post PF-03654746/placebo dose at each intervention period and (for congestion only) 3 hrs 40 min post PF-03654746/placebo dose (Post-oxymetazoline) at each intervention period.
Time Frame: 2 hrs 10 min, 2 hrs 25 min, 2 hrs 40 min post dose (Pre-allergen challenge); 2 hrs 55 min, 3 hrs 10 min, 3 hrs 25 min post dose (Post-allergen challenge); 3 hrs 40 min post dose (Post-oxymetazoline) on Day 1 of each intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Number analyzed (Participants) | 20 | 19 | 19 | 19
units on a scale
  Nasal congestion: Pre-allergen challenge | 0.2 (0.36) | 0.4 (0.42) | 0.4 (0.57) | 0.4 (0.59)
  Nasal congestion: Post-allergen challenge | 1.5 (1.20) | 1.8 (1.30) | 1.9 (1.42) | 2.2 (1.48)
  Nasal congestion: Post-oxymetazoline | 0.8 (1.16) | 0.8 (1.21) | 0.9 (0.85) | 0.9 (1.20)
  Nasal Itching: Pre-allergen challenge | 0.0 (0.07) | 0.1 (0.23) | 0.0 (0.08) | 0.1 (0.31)
  Nasal Itching: Post-allergen challenge | 0.4 (0.71) | 0.8 (1.10) | 0.9 (1.12) | 1.4 (1.43)
  Rhinorrhea: Pre-allergen challenge | 0.1 (0.23) | 0.1 (0.17) | 0.2 (0.39) | 0.1 (0.33)
  Rhinorrhea: Post-allergen challenge | 0.6 (1.01) | 1.1 (1.48) | 1.3 (1.30) | 1.9 (1.42)
Statistical Analysis 1: Comparison: PF-03654746 10 mg vs Placebo; Nasal congestion: An ANOVA mixed model was assessed with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.011, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 2: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.127, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 3: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.103, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 4: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.218, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.905, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.273, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 7: Comparison: PF-03654746 10 mg vs Placebo; Nasal Itching: An ANOVA mixed model was assessed with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.000, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 8: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.055, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 9: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.012, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 10: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.048, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 11: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.496, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 12: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 5, analysis 7]; Test type: Superiority or Other; p = 0.190, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 13: Comparison: PF-03654746 10 mg vs Placebo; Rhinorrhea: An ANOVA mixed model was assessed with sequence, period and treatment as fixed effects and participant within sequence as a random effect; Test type: Superiority or Other; p = 0.000, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 14: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.019, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 15: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.009, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 16: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.061, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 17: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.778, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 18: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 5, analysis 13]; Test type: Superiority or Other; p = 0.102, ANOVA — [p-value comment as in outcome 1, analysis 4]

6. Secondary Outcome: Nasal Symptom Scores: Sneezing
Description: The absolute number of sneezes was recorded by the participants under supervision of study personnel. Nasal symptom score for sneezing was assessed as the total number of sneezes of each intervention period at specified time-points for the post-diluent and post-challenge and post where 'post-diluent, pre-allergen challenge' included 2 hrs 10 min, 2 hrs 25 min and 2 hrs 40 min post PF-03654746/placebo dose at each intervention period and 'post-allergen challenge' included 2 hrs 55 min, 3 hrs 10 min and 3 hrs 25 min post PF-03654746/placebo dose at each intervention period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: sneezes
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Number analyzed (Participants) | 20 | 19 | 19 | 19
sneezes
  Sneezing: Pre-allergen challenge | 0.0 (0.07) | 0.1 (0.23) | 0.1 (0.61) | 0.1 (0.17)
  Sneezing: Post-allergen challenge | 0.7 (1.54) | 0.6 (0.92) | 1.2 (1.94) | 3.6 (3.24)
Statistical Analysis 1: Comparison: PF-03654746 10 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.000, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 2: Comparison: Allegra-D vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.000, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 3: Comparison: PF-03654746 1 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.000, ANOVA — P-value was based on a one-sided test. There were no further adjustments for multiplicity
Statistical Analysis 4: Comparison: PF-03654746 10 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.217, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 5: Comparison: PF-03654746 1 mg vs Allegra-D; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.156, ANOVA — [p-value comment as in outcome 1, analysis 4]
Statistical Analysis 6: Comparison: PF-03654746 10 mg vs PF-03654746 1 mg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.848, ANOVA — [p-value comment as in outcome 1, analysis 4]

7. Other Pre Specified Outcome: Serum PF-03654746 Concentration
Description: Only participants receiving PF-03654746 were analyzed for this outcome measure. Mean serum concentration of PF-03654746 was calculated of each intervention period.
Time Frame: 1 hr 30 min post dose on Day 1 of each intervention period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg
Number analyzed (Participants) | 20 | 19
nanogram per milliliter (ng/mL) | 34.16 (17.85) | 2.78 (1.55)

ADVERSE EVENTS:
Description: All participants included in safety analysis set were evaluable for adverse events. Participants at risk = 20, 19, 19, 19 for each arm group, respectively.
Arm/Group | PF-03654746 10 mg | PF-03654746 1 mg | Allegra-D | Placebo
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 5/20 | 2/19 | 0/19 | 2/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-03654746 10 mg (N=20) | PF-03654746 1 mg (N=19) | Allegra-D (N=19) | Placebo (N=19)
Feeling jittery (General disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.